CLINICAL TRIAL: NCT03409978
Title: Feasibility of a Smartphone Application for Computer-based Movement Analysis During the Fidgety Period of General Movements
Brief Title: Smartphone App for Analysis of General Movements in Young Infants
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University of Illinois at Chicago (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Christian Medical College, Vellore, India (Other); University Ghent (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/913
Record Dates: First submitted 2018-01-10; First posted 2018-01-25 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: Infants, newborn; General Movements; Video Recording; Mobile Applications; Prognosis; Parents
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-Motion app for movement analysis: Participants will be recruited from infants referred to the high-risk follow-up clinic at the hospital. These at-risk children are included in the regular clinical follow-up program comprising a standard examination at 3 months corrected age (fidgety general movements period). Infant/families from St. Olavs Hospital (n= 15), in Norway, Lurie Children's Hospital (n=15), Chicago, USA, Christian Medical College (n=15), Vellore, India, University of Ghent (n=15), Belgium, and Hillerød Hospital (n=30), Copenhagen, Denmark will be invited to participate.
  Interventions: Device: in-Motion app

INTERVENTIONS:
Device: in-Motion app — mobile phone application for recording fidgety movements at home

SUMMARY:
Analysis of spontaneous movements in young infants from video recordings is recommended as an early medical assessment tool for prediction of cerebral palsy in high-risk infants. Such video recording have previously been performed in follow-up programs at hospitals using semi standardized video set-ups. The research group behind this study develops a smart-phone application that makes it possible for parents to video film their infant spontaneous movements at home, upload and send the video for analysis at the hospital provided by experts. The objectives of the study are to assess the feasibility of the In-Motion app for video recording of infant spontaneous movements, upload and send the video to St. Olavs Hospital in Trondheim, Norway, for assessment, and how parents experience this. 90-120 high-risk infants from Norway, Denmark, Belgium, USA, Great Britain and India will participate. Parents will record their infant spontaneous movements and answer questionnaires. Video quality will be evaluated by experts within the field and their use for computer-based assessment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infants referred to high-risk follow-up at the hospital

Exclusion Criteria:

* Unstable medical condition, progressive disorders, or diagnosis with a specific syndrome affecting motor development.

Ages: 12 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: High-risk infants included in the regular clinical follow-up program comprising a standard examination at 3 months corrected age.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of recordings that movement video recordings fulfil requirements needed for observation and classification of fidgety general movements | 17 weeks post term age
Ease of use of the In-Motion App in score on the Software usability scale (SUS) as part of a questionnaire sent to users two weeks after received video recordings | 2 weeks after received video recordings
  SUS is a 10 item questionnaire with 5 response options between 'strongly disagree' and 'strongly agree'. All values are scaled from 0 to 4 (with four being the most positive response). The range of possible values is converted from 0 to 100. A SUS score above a 68 would be considered above average. See https://measuringu.com/sus/
Correlation between computer-based software estimates by smartphone videos performed by parents at home and standard videos performed at the hospital follow-up clinic | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Adde, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (3):
- Ghent University, Ghent, Belgium
- Hillerød Hospital, Copenhagen, Denmark
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Adde L, Brown A, van den Broeck C, DeCoen K, Eriksen BH, Fjortoft T, Groos D, Ihlen EAF, Osland S, Pascal A, Paulsen H, Skog OM, Sivertsen W, Stoen R. In-Motion-App for remote General Movement Assessment: a multi-site observational study. BMJ Open. 2021 Mar 4;11(3):e042147. doi: 10.1136/bmjopen-2020-042147. PMID 33664072